CLINICAL TRIAL: NCT04023162
Title: Controlled, Randomized, Blind Trial Therapy Exercises and Operant Conditioning for Chronic Nonspecific Low Back Pain
Brief Title: Therapy Exercises and Physiotherapy Delivered Operant Conditioning in the Treatment Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antonija Hrkać (Other)
Responsible Party: Sponsor-Investigator, Antonija Hrkać, Master of Physiotherapy, Postgraduate Study in Health Sciences, University of Mostar
Organization: University of Mostar (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Studija I
Record Dates: First submitted 2019-07-14; First posted 2019-07-17 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2019-07

CONDITIONS: Chronic Nonspecific Low Back Pain
Keywords: Low Back Pain; Nonspecific; Operant Conditioning; Graded Activity; Therapy Exercise
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: By randomization, the participants will be divided into three groups, two experimental groups, and a control group. In the first experimental group, the investigated interventions will consist of Therapy Exercise and Back School. In the second experimental group, in addition to the Therapy Exercise and the Back School, operative conditioning will be performed by the master of physiotherapy. The participants in the control group will be exposed to the usual treatment.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of interventions that will be applied in this study, blinding of therapists who will carry out the intervention regarding Therapy Exercise will not be possible to implement, but physiotherapists (apart from the study designer) will not know the study hypothesis. Fully blinding of the examinees is also impossible to implement, but partially blinding will occur, as the participants in the Graded Activity group will not explain the applied behavioral therapy. Blinding will be applied to researchers who will collect data (measure outcomes) and statisticians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biomedical (Physiotherapy) group (Experimental): Therapy Exercise and Back School; 8 sessions during 4 weeks (2 times a week), with one session lasting 60 min.
  Interventions: Behavioral: Group-based Therapy Exercise; Behavioral: Back School
- Biopsychosocial (Graded Activity) group (Experimental): Operant Conditioning implement in Physiotherapy, Therapy Exercises and Back School; 8 sessions during 4 weeks (2 times a week), with one session lasting 60 min.
  Interventions: Behavioral: Graded Activity; Behavioral: Group-based Therapy Exercise; Behavioral: Back School
- Usual care (No Intervention): Usual care and written instructions on Therapy Exercise and Back School for self-care.

INTERVENTIONS:
Behavioral: Graded Activity — Active participation of participants, Overcoming and eliminating negative behaviors, Encouraging positive behavior in pain, Overcoming the fear of the movement, Motivation to implementation pre-set specific goals.
  Other Names: Physiotherapy - Provided Operant Conditioning
  Arms: Biopsychosocial (Graded Activity) group
Behavioral: Group-based Therapy Exercise — Aerobic exercise, Stretching exercise and flexibility, Range of motion, Balance and coordination, Breathing exercises Stabilization exercise Muscle strength training exercise
  Other Names: Exercises Therapy, Kinesitherapy
  Arms: Biomedical (Physiotherapy) group; Biopsychosocial (Graded Activity) group
Behavioral: Back School — Basic information of Low Back Pain - anatomy, physiology, causes, treatment. Correct postures - standing, sitting, driving, sleeping, Correct body movements - lifting, pushing, walking.
  Arms: Biomedical (Physiotherapy) group; Biopsychosocial (Graded Activity) group

SUMMARY:
This study investigates the effect of two physiotherapy models in the treatment of chronic nonspecific low back pain. Participants will be divided into three groups, two experimental and one control. In both experimental groups, the participants will be included in the intensive program of Therapy Exercises, under the supervision and guidance of the physiotherapist, and the group will differ in implemented behavioral therapy (which he will implement by a physiotherapist). In the control group, subjects will receive the usual treatment. The Back School will be applied in all groups.

DETAILED DESCRIPTION:
Low back pain is a global public health problem, one of the main causes of disability of the population, as well as enormous economic costs in the health system. This claim specifically relates to chronic low back pain. The clinical picture of chronic low back pain in addition to pain, muscle spasm, and functional disability dominate psychological problems, which significantly affect the outcome of treatment. The multidisciplinary approach to the treatment of chronic low back pain has proven to be the most effective, bad economically unacceptable, and unavailable in many countries. Therefore, it is necessary to find the most effective and economically most acceptable approach to the treatment of chronic low back pain.

Physiotherapy is an unavoidable method of treating this painful condition, and changes in treatment approaches are most evident in this medical profession. Recently, physiotherapy includes two models in the treatment of chronic low back pain. A biomedical model consisting of well-known physiotherapy methods and a Biopsychosocial model that, in addition to known physiotherapy methods, includes a part of cognitive-behavioral therapy associated with motion and behavior, operative conditioning. Therapy exercise is an effective method indispensable part of both models of physiotherapy.

The reason for changes in physiotherapy is a varied clinical picture of chronic low back pain. Evidence-based effectiveness of therapy exercise has been determined on reduction of the body's symptoms, pain, and functional disabilities. The effect of reducing psychological symptoms has been poorly investigated. Also, the use of therapeutic exercises in the practice creates several concerns related to the intensity of exercise, mode and time-frame of their application, and the type or method of exercise.

Because it's already a known effect of operant conditioning through a multidisciplinary approach to reducing the psychological symptoms of chronic low back pain, it is suggested that this part of cognitive-behavioral therapy be implemented in physiotherapy, namely therapy exercise. Studies aimed to determine the effect of biopsychosocial physiotherapy models are scarce and insufficiently clear.

The aims of this study are:

1. Determine the effectiveness of a biomedical model of physiotherapy in the treatment of chronic nonspecific low back pain,
2. Determine the effectiveness of the biopsychosocial model of physiotherapy in the treatment of chronic nonspecific low back pain, and
3. Compare the effectiveness of these interventions.

ELIGIBILITY:
Inclusion Criteria:

* People with a diagnosis of nonspecific pain in the spinal area with symptoms of pain 3 and > months, confirmed by a doctor specialist family medicine,
* Age from 18 to 75 years of life,
* Both sexes.

Exclusion Criteria:

* Acute and Subacute low back pain,
* Specific Low Back Pain,
* Operative interventions on the spine,
* Other health problems of the patient: pregnancy or gynecological diseases, blood vessels, elevated blood pressure, malignant and benign tumors in the spine, spinal abnormalities, spinal traumas, urological disorders and psychological disorders,
* Mental health problems that prevent the verbal expression and understanding of the questionnaire, and
* People who have been included in the therapeutic exercise program for the past 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) Pain Score | Baseline, 4 week (post-treatment), 3 month i 6 month post-randomization
  Self-reported pain intensity, Each item scored 0-100 mm (0=No pain; 100=Pain as bad as can be).

SECONDARY OUTCOMES:
Change in Roland Morris Disability Questionnaire (RMDQ) Score | Baseline, 4 week (post-treatment), 3 month i 6 month post-randomization
  Self-reported assessment of functional disability in low back pain. It consists of 24 questions that question how crossbreeding affects daily activities, and is calculated by a sum of total answers of 0 to 24. A larger sum indicates greater disability.
Change in Goniometry of spine (ROM) Score | Baseline, 4 week (post-treatment), 3 month i 6 month post-randomization
  Functional assessment of range of motion in lumbal spine with goniometer - flexion, extension and latero-flexion right and left;
Change in Finger to Floor Test (FTF) | Baseline, 4 week (post-treatment), 3 month i 6 month post-randomization
  Functional assessment of lumbar spine flexion; with a centimeters band the distance between the middle finger and the floor is measured.
Change in Prone Double Straight Leg Raise Test (PDSLRT) Score | Baseline, 4 week (post-treatment), 3 month i 6 month post-randomization
  Assessment of muscle strength back extensors, measures are in seconds.
Change in Hospital Anxiety and Depression Scale (HAD) Score | Baseline, 4 week (post-treatment), 3 month i 6 month post-randomization
  Self-assessment intensity of depression and anxiety. It consists of 14 questions, 7 questions for assessing depression and 7 for assessing anxiety. Responses are scored at four levels from 0 to 3 (0 = not at all, 3 = all the time) so the results may vary from 0 to 21 for depression or anxiety. Respondents with scores 0-7 are not depressed/anxious, 8-10 indicate a marginal state and 11-21 represent depression/anxiety.
Change in Fear-Avoidance Beliefs Questionnaire (FABQ) Score | Baseline, 4 week (post-treatment), 3 month i 6 month post-randomization
  Assessment to avoid movement due to fear of pain. It consists of 16 particles and each question is evaluated from 0 to 6. A higher score indicates a greater presence of fear/avoidance. FABQ is divided into two parts (work and physical activity), one measures the correlation of work with the current feeling of pain in low back pain, and the second connection of physical activity on the current sense of pain in low back pain.
Change in Short Form Health Survey 12 (SF-12) core | Baseline, 4 week (post-treatment), 3 month i 6 month post-randomization
  Questionnaire of assessment quality of life. The instrument by which the subjective sense of individual health is measured through 12 questions examines the physical, psychological, and social consequences caused by impaired health. With this questionnaire, it is possible to quantitatively compare each dimension of health, because the score for each question is transformed into standard values and placed on the scale from 0 to 100 (the higher the score the better health) and thus get two major dimensions of health: physical (Physical Common Score-PCS)and mental health (Mental Common Score-MCS).
Questionnaire assessment of satisfaction with treatment | 6 month post-randomization
  The assessment of satisfaction with interventions as well as cost-effectiveness was measured using single questions and answers on the 5-item Likert scale, from completely dissatisfied to completely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Antonija Hrkać, Principal Investigator — Faculty of Health Science
Locations (2):
- Bosnia and Herzegovina (2):
  - Dom zdravlja Mostar, Mostar
  - Rehabilitacijski centar "Život", Mostar

IPD SHARING:
Plan to Share IPD: Yes
All of individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Background] Ma VY, Chan L, Carruthers KJ. Incidence, prevalence, costs, and impact on disability of common conditions requiring rehabilitation in the United States: stroke, spinal cord injury, traumatic brain injury, multiple sclerosis, osteoarthritis, rheumatoid arthritis, limb loss, and back pain. Arch Phys Med Rehabil. 2014 May;95(5):986-995.e1. doi: 10.1016/j.apmr.2013.10.032. Epub 2014 Jan 21. PMID 24462839
- [Background] Wong JJ, Cote P, Sutton DA, Randhawa K, Yu H, Varatharajan S, Goldgrub R, Nordin M, Gross DP, Shearer HM, Carroll LJ, Stern PJ, Ameis A, Southerst D, Mior S, Stupar M, Varatharajan T, Taylor-Vaisey A. Clinical practice guidelines for the noninvasive management of low back pain: A systematic review by the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration. Eur J Pain. 2017 Feb;21(2):201-216. doi: 10.1002/ejp.931. Epub 2016 Oct 6. PMID 27712027
- [Background] Henschke N, Ostelo RW, van Tulder MW, Vlaeyen JW, Morley S, Assendelft WJ, Main CJ. Behavioural treatment for chronic low-back pain. Cochrane Database Syst Rev. 2010 Jul 7;2010(7):CD002014. doi: 10.1002/14651858.CD002014.pub3. PMID 20614428
- [Background] Hall A, Richmond H, Copsey B, Hansen Z, Williamson E, Jones G, Fordham B, Cooper Z, Lamb S. Physiotherapist-delivered cognitive-behavioural interventions are effective for low back pain, but can they be replicated in clinical practice? A systematic review. Disabil Rehabil. 2018 Jan;40(1):1-9. doi: 10.1080/09638288.2016.1236155. Epub 2016 Nov 21. PMID 27871193
- [Background] Lamb SE, Hansen Z, Lall R, Castelnuovo E, Withers EJ, Nichols V, Potter R, Underwood MR; Back Skills Training Trial investigators. Group cognitive behavioural treatment for low-back pain in primary care: a randomised controlled trial and cost-effectiveness analysis. Lancet. 2010 Mar 13;375(9718):916-23. doi: 10.1016/S0140-6736(09)62164-4. Epub 2010 Feb 25. PMID 20189241
- [Background] Gordon R, Bloxham S. A Systematic Review of the Effects of Exercise and Physical Activity on Non-Specific Chronic Low Back Pain. Healthcare (Basel). 2016 Apr 25;4(2):22. doi: 10.3390/healthcare4020022. PMID 27417610
- [Background] National Collaborating Centre for Primary Care (UK). Low Back Pain: Early Management of Persistent Non-specific Low Back Pain [Internet]. London: Royal College of General Practitioners (UK); 2009 May. Available from http://www.ncbi.nlm.nih.gov/books/NBK11702/ PMID 20704057
- [Background] Searle A, Spink M, Ho A, Chuter V. Exercise interventions for the treatment of chronic low back pain: a systematic review and meta-analysis of randomised controlled trials. Clin Rehabil. 2015 Dec;29(12):1155-67. doi: 10.1177/0269215515570379. Epub 2015 Feb 13. PMID 25681408
- [Result] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Derived] Hrkac A, Bilic D, Cerny-Obrdalj E, Baketaric I, Puljak L. Comparison of supervised exercise therapy with or without biopsychosocial approach for chronic nonspecific low back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Nov 8;23(1):966. doi: 10.1186/s12891-022-05908-3. PMID 36348309